CLINICAL TRIAL: NCT05980559
Title: Evaluation of Botulinum Toxin Injection in Treatment of Bruxism
Brief Title: Evaluation of BTX Injections in Treatment of Bruxism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Walaa Ali Elwakil, Lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Botulinum toxin in bruxism
Record Dates: First submitted 2023-06-22; First posted 2023-08-08 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Bruxism
Keywords: Botulinum toxin; Electromyographic; occlusense
MeSH Terms: conditions — Bruxism | interventions — incobotulinumtoxinA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One Group (Experimental): Patients will be injected with 50 MU of botulinum toxin and Surface qualitative Electromyography, maximum bite force and visual pain scale will be taken before and after 1, 3 months
  Interventions: Drug: Xeomin

INTERVENTIONS:
Drug: Xeomin — 50 units of Incobotulinumtoxin A (BTX A) Xeomin® Injections into the masseter and temporalis muscles bilaterally (15 Units per muscle applied with 2 injections in each masseter muscle) (10 Units per muscle applied with 2 injections in each temporalis muscle)

SUMMARY:
Aim of this study is to evaluate the effect of botulinum toxin type A (Xeomin®) on patients complaining from bruxism.

The study will be a one arm clinical trial. Twelve subjects reporting bruxism irresponsive to conventional treatment modalities will be recruited and will be injected with botulinum toxin A (Xeomin®) in both masseter and temporalis muscles. Pain levels, Electromyographic activity and maximum occlusal force will be recorded in the subjects before injection and at 1 and 3 months after injection to determine the effect of treatment

DETAILED DESCRIPTION:
Bruxism is a parafunctional activity of the masticatory muscles, characterized by jaw clenching and/or tooth grinding. It was suggested in international consensus conference that bruxism should have two distinct definitions. Sleep bruxism is a muscular action, either rhythmic or not, that takes place while sleeping, and an Awake bruxism which is a muscle disorder characterized by repeated or prolonged teeth contact with clenching of the jaw.

Bruxism is a highly prevalent condition. More than 85% of the general population admit to bruxism at some time during their life. According to reports, the prevalence of awake bruxism is about 24% in the adult population, while the prevalence of bruxism when sleeping is estimated to be around 16% of the same population.

The three muscles that responsible for the jaw closure and the majority of the biting force is the masseter, temporalis, and medial pterygoid muscles. About 43% of the intrinsic strength of jaw closure comes from the masseter, 36% from the temporalis, and 21% from the medial pterygoid.

The diagnosis of bruxism is made on the basis of self-reporting of clenching or grinding the teeth, as well as evaluating tooth mobility, tooth wear, bruxism-related sounds, or jaw muscle pain and other clinical findings of the temporo-mandibular joint (TMJ).

Bruxism has been noted in dentistry as a risk factor for tooth fracture and dental prosthesis damage, periodontal disease and possibly pain in the teeth, jaw, masticatory muscles, and temporo-mandibular joint. The etiology and pathophysiology of bruxism are still unknown, despite several potential causes have been suggested, including emotional stress, neurological diseases, specific medications, and occlusal interferences.

Physical therapy, occlusal splints, and pharmacological management have all been investigated as potential treatment modalities for bruxism, but they have not been proven to be completely effective because they mostly treat patients' symptoms and signs rather than treating the underlying cause of the condition. These treatment modalities helped only in limiting the damaging effects of bruxism on the anatomical structures.

Irreversible occlusal correction has been found ineffective and it is not supported by the available research. Occlusal splints have been applied to prevent overloading the temporomandibular joint elements and muscles of the jaw in addition to prevent tooth attrition. The efficacy of occlusal splints has given conflicting results.

Botulinum toxin (Botox) is currently known to be a useful treatment for a wide range of neurological conditions, and it is used for its therapeutic and cosmetic effect. It is formed by the anaerobic bacterium Clostridium botulinum and has paralytic properties as it can inhibit acetylcholine release, which can ultimately inhibit muscle contraction. Botulinum toxin comes in seven forms : A, B, C, D, E, F, and G. Type A, which cleaves the plasma protein SNAP-25, is the most commonly used commercially and clinically. It is injected intramuscularly, and its effect lasts between three and six months and this transient denervation depends on the dose and volume of toxin.

Since bruxism is caused by involuntary spasms of the jaw muscles, botulinum toxin has been experimented; initial results show that it is safe and effective. The injections generally take one week to start working and two weeks for a full effect, which lasts on average three to six months, and slowly wears off.

The purpose of this study is to evaluate the efficacy of injecting botulinum toxin A into the masseter muscle in participants with bruxism, using a pain scale, Electromyography and occlusense device.

The null hypothesis tested in this study is that there will be no significant difference in the pain level, muscles contractility and biting forces in patients injected with botulinum toxin

ELIGIBILITY:
Inclusion Criteria:

1. Patient between 20 and 60 years of age.
2. Pain related to the masseter muscles and TMJ area due to bruxism.
3. Patient who has never received botulinum toxins.
4. Patient who did not respond to the conventional treatments (analgesic, physiotherapy, relaxation technique and maxillary retainer).

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Neuromuscular diseases, including neurogenic impairment of the face and patients with underlying neurological disorders.
3. Patients with epilepsy or a previous seizure episode.
4. Injection site infection (masseter or temporalis).
5. Hypersensitivity or allergy to botulinum toxin or any of its excipients.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in electromyographic activity of temporalis and masseter muscles bilaterally. | Assessment will be done before the injection versus 1 and 3 months after injection
  Analyze the electromyographic activity of temporalis and masseter muscles bilaterally. The acquisitions will be performed twice with the rest position of the mandible (RPM) for 10 seconds, in maximal intercuspal position for 5 seconds, and maximal teeth clenching with 10-mm thick cotton rolls between the posterior teeth for 5 seconds, bilaterally, and the median of values will be obtained. The unit of measurement used in the Electromyographic records will be microvolts (μV).

SECONDARY OUTCOMES:
Change in Pain Assessment | Assessment will be done before the injection versus 1 and 3 months after injection
  The pain will be measured using a visual analogue scale (VAS). The patient will be asked to mark on a line that measured 100 mm in length where she/he reflected her/his perceived pain. The scores of the scale will be determined by measuring the distance in mm from the beginning to the point indicated by the patient (point (0): no pain and point (100): the highest levels of pain).
Change in maximum bite force | Assessment will be done before the injection versus 1 and 3 months after injection
  Computerized occlusal analysis will be conducted using the Occlusense device to record and analyze the biting force of each patient. The system use a 100-µm thick recording sensor. All scanning procedures will be carried out by the same clinician and at the same time of the day to avoid variability. The size of the sensor, large or small, will be chosen to suit the patient's dental arch. Prior to any occlusal acquisition sensitivity of the device will be adjusted. The patient will be asked to bite on the sensor, and a record for the maximum biting force on the first molar region (key of occlusion).
Change in Bruxism symptom questionnaire | questionnaire will be done before the injection versus 1 and 3 months after injection
  to evaluate the subjective bruxism symptoms consisted of three items: (1) How often do you think that you had bruxed at night during the past 1 month? (2) How often have you heard from your sleeping partner that you bruxed during the past 1 month? (3) How often during the past month have you felt jaw stiffness on waking? The responses to each item were based on a 0-5 scale where 0 = none, 1 = very seldom, 2 = seldom, 3 = often (half the mornings), 4 very often, 5 = every day. The rationale was that previous reports have used subjective measures, and we wished to compare our results with the previous data.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab S. Hassan, Professor, Study Director — Alexandria University; Gaafar N. Elhalawani, Lecturer, Study Chair — Alexandria University; Walaa A. Elwakil, Lecturer, Study Chair — University of Alexandria; Marwa M. Mancy, Bachelors, Principal Investigator — Alexandria University